CLINICAL TRIAL: NCT04192747
Title: Evaluation of a Sirolimus Eluting Bioadaptor as Compared to a Zotarolimus Eluting Stent in De Novo Native Coronary Arteries ELX-CL-1805
Brief Title: The Elixir Bioadaptor vs. The Onyx Stent in De Novo Native Coronary Arteries
Acronym: BIOADAPTOR RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELX-CL-1805
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Disease; Coronary Stenosis
Keywords: Coronary Ste; Bioadaptor; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Single-blind, 1:1 Randomized trial of parallel design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Elixir Bioadaptor (ELX1805J) (Experimental): The Elixir Bioadaptor (ELX1805J) 2.25 - 4.0 mm diameter and 14,15,18, 23, 28, 32 and 38 mm in length
  Interventions: Device: Percutaneous Coronary Intervention
- Medtronic Resolute Onyx Stent (Active Comparator): The Medtronic Resolute Onyx Stent 2.25 - 4.0 mm diameter and 15, 18, 22, 30, 34 and 38 mm in length
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Percutaneous coronary intervention of de novo native coronary artery lesions

SUMMARY:
The objective of this study is to verify the safety and efficacy of the investigational device (ELX1805J) for the treatment of ischemic heart disease due to de novo, native coronary artery lesions

DETAILED DESCRIPTION:
The Bioadaptor RCT Study is a prospective, 1:1 randomized study of parallel designed, that will enroll up to 444 patients requiring treatment of up to two de novo coronary lesions of ≤ 34 mm in length in vessels of ≥ 2.25 mm and ≤ 4.0 mm in diameter.

One or two designated target lesions, located in separate epicardial vessels (RCA, LCX or LAD), and meeting the inclusion/exclusion criteria may be treated with the ELX1805J (DynamX Bioadaptor) or Resolute Onyx stent

The primary safety endpoint is Target Lesion Failure (TLF) at 12 months. TLF is a composite endpoint defined as cardiac death, target vessel MI, and clinically-indicated target lesion revascularization

Additional secondary safety and effectiveness endpoints will be evaluated at 30 days, 6 and 12 months and 2-5 years.

Using visual assessment, the target lesion must measure ≥ 2.25 mm and ≤ 4.0 mm in diameter and ≤ 34 mm in length able to be covered by a single ELX1805J or Resolute Onyx stent including 2 mm of healthy vessel on either side of the planned treatment area.

The patient will be eligible for device implantation only after satisfactory lesion pre-dilatation defined as: ≥ TIMI 2 flow, and no dissection greater than Grade B (NHLBI) able to be covered with a single device

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

Patients who meet all of the following criteria are eligible:

1. Patient must be ≥ 20 years of age.
2. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
3. Patients who are able to take dual anti-platelet therapy for 1 year following the index procedure and anticoagulants prior to/during the index procedure.
4. The subject is an acceptable candidate for Percutaneous Transluminal Coronary Angioplasty (PTCA), stenting, and emergent Coronary Artery Bypass Graft (CABG) surgery.
5. The subject or subject's legally authorized representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board or Ethics Committee of the respective clinical site.
6. Women of childbearing potential with a negative pregnancy test within 7 days and women who are not pregnant or nursing
7. Patient must agree to undergo all clinical study required follow up visits, angiograms, and imaging testing
8. Patient must agree not to participate in any other clinical research study for a period of one year following the index procedure
9. Target lesion(s) must be de novo and located in a native coronary artery with a vessel mean diameter of ≥ 2.25 and ≤ 4.0 mm.
10. Target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of > 1. When two target lesions are treated, they must be located in separate major epicardial vessels
11. visually estimated target lesion length is ≤ 34mm mm and must be able to be covered by a single 14/15/18/23/28/32/38 mm ELX1805J stent and have at least 2 mm of healthy vessel on either side Or
12. The visually estimated target lesion length is ≤ 34mm mm and must be able to be covered by a single 15/18/22/30/34/38 mm ZES stent respectively and have at least 2 mm of healthy vessel on either side.
13. The lesion(s) must be successfully pre-dilated prior to enrollment Mandatory pre-dilatation includes the use of 2 orthogonal views to confirm lesion inclusion and exclusion criteria and successful pre-dilatation defined as balloon inflation without waist and a lumen diameter no less than 0.5 mm smaller than the vessel diameter.
14. Percutaneous intervention of lesions in a non-target vessel if:

    * Not part of a another clinical investigation
    * ≥ 30 days prior to the study index procedure
    * ≥ 6 months after the study index procedure (planned)
15. Percutaneous intervention of lesions located in the target vessel if:

    * Not part of a clinical investigation
    * ≥ 6 months prior to the study index procedure
    * >12 months after the study index procedure (planned)
    * Previous intervention was distal to and >10 mm from the target lesion

Exclusion Criteria:

1. The patient was diagnosed with an acute myocardial infarction within the past 72 hours and the CK and CKMB have not returned to normal (or cTn >15x ULN) and the patient is experiencing clinical symptoms indicative of ongoing ischemia
2. Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, prasugrel or ticagrelor, cobalt, nickel, chromium, molybdenum, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
3. Patients with a history of allergic reaction or serious hypersensitivity to drugs exhibiting interactions with sirolimus, zotarolimus, everolimus, tacrolimus, temsirolimus, biolimus and other rapamycin, derivatives or analogues) or similar drugs
4. Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel or other P2Y12 inhibitors.
5. Patient presenting with chronic (permanent) atrial or ventricular arrhythmia or current unstable ventricular arrhythmias
6. Patient has a known left ventricular ejection fraction (LVEF) < 30%
7. Patient has received a heart or other organ transplant or is on a waiting list for any organ transplant
8. Patient has a malignancy that is not in remission.
9. Patient is receiving immunosuppression therapy other than steroids and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
10. Patient is receiving chronic anticoagulation therapy (e.g., heparin, coumadin) that cannot be stopped and restarted according to local hospital standard procedures.
11. Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected to have cirrhosis of Child-Pugh ≥ Class B within 7 days before study procedure
12. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL within 7 days before study procedure, or patient on dialysis)
13. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
14. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
15. Patient has had a significant GI or urinary bleed within the past six months
16. Patient has severe symptomatic heart failure (i.e., NYHA class IV)
17. Patient has a medical condition that precludes safe 6 French sheath insertion
18. Patient has other medical illness or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
19. Patient is already participating in another clinical research study which has not reached the primary endpoint (long-term follow-up is not an exclusion)
20. Other patients whom primary investigator or subinvestigator determined to be ineligible for this clinical study
21. Patients with bypass graft to the target vessel or lesion is located in a bypass graft
22. Patients with stent implanted within 10 mm of proximal or distal end of target lesion
23. Patients with a target lesion involving a bifurcation of which the side branch will be jailed by the struts and:

    * Side branch ≥ 2.5 mm in diameter,
    * Side branch requiring predilatation (including Kissing Balloon Technique), or
    * Side branch has an ostial lesion or lesion with > 50% stenosis
24. Patients suspected or confirmed with the QCA analysis of having stenotic lesion of more than 50% in target vessel in addition to target lesion
25. Patients with target lesion in ostia located within 5 mm of origin of LAD, LCX or RCA
26. Patients with stenotic lesion in left main trunk
27. Patients with target lesion that is a chronic total occlusion (CTO) or ≤ TIMI 1 coronary flow in the target vessel
28. Patients with target vessel that contains thrombus as indicated in pre-procedure angiographic, IVUS or OCT images
29. Excessive tortuosity ≥ two 45° angles or extreme angulation (≥ 90°) proximal to or within the target lesion
30. Patients with target vessel that has moderate to severe calcification that prevents complete angioplasty balloon (POBA with non-compliant balloon, or scoring balloon,) inflation or requires other devices such as rotational atherectomy, rotoblator.
31. Patients with dissection of Grade A or B that cannot be covered (including 2mm distal to the dissection) with a single study device or with dissection of Grade C or higher
32. Patients with 2 or more target lesions on 1 branch or target lesions on 3 branches that need to be treated during study procedure
33. Target lesion involves a myocardial bridge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2027-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Chief Director, Shonan Kamakura General Hospital
Locations (36):
- Belgium (4):
  - AZ Middelheim Hospital, Antwerp
  - AZ Sint Jan Brugge, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Universitaire Ziekenhuizen Leuven, Leuven
- Germany (12):
  - Kerkhoff Klinik GmbH, Bad Nauheim
  - Segeberger Kliniken GmbH, Bad Segeberg
  - REGIOMED Klinikum Coburg, Coburg
  - St. Johannes Hospital, Dortmund
  - Universitatsklinikum Erlangen, Erlangen
  - Elisabeth Krankenhaus Essen, Essen
  - MVZ CCB Frankfurt, Frankfurt
  - Universitatsklinikun Giessen, Giessen
  - Universitätsklinikum Jena, Jena
  - UKSH Kiel Klinik, Kiel
  - Universitätsmedizin-Mainz, Mainz
  - Krankenhaus der barmherzigen Bruder, Trier
- Japan (14):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Shinkoga Hospital, Kurume, Fukuoka
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Takahashi Hospital, Tsuchiura, Ibaraki
  - Tsuchiura Kyodo Hospital, Tsuchiura, Ibaraki
  - Tenyokai Central Hospital, Kagoshima, Kagoshima-ken
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kanto Rosai Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City Eastern Hospital, Yokohama, Kanagawa
  - Kumamoto Rousai Hospital, Kumamoto, Kumamoto
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Oumi Hachiman City General Medical Center, Hachiman, Shiga
  - Cardiovascular Reaearch Institute, Tokyo
  - Teikyo University Hospital, Tokyo
- New Zealand (6):
  - Auckland City Hospital, Auckland
  - Middlemore Clinical Trials Trust, Auckland
  - Waikato Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - North Shore Hospital, Takapuna

REFERENCES:
- [Derived] Saito S, Bennett J, Nef HM, Webster M, Namiki A, Takahashi A, Kakuta T, Yamazaki S, Shibata Y, Scott D, Vrolix M, Menon M, Mollmann H, Werner N, Neylon A, Mehmedbegovic Z, Smits PC, Morice MC, Verheye S; BIOADAPTOR-RCT Collaborators. Percutaneous Coronary Treatment With Bioadaptor Implant vs Drug-Eluting Stent: 2-Year Outcomes From BIOADAPTOR RCT. JACC Cardiovasc Interv. 2025 Apr 28;18(8):988-997. doi: 10.1016/j.jcin.2025.01.426. Epub 2025 Feb 26. PMID 40057888
- [Derived] Saito S, Bennett J, Nef HM, Webster M, Namiki A, Takahashi A, Kakuta T, Yamazaki S, Shibata Y, Scott D, Vrolix M, Menon M, Mollmann H, Werner N, Neylon A, Mehmedbegovic Z, Smits PC, Morice MC, Verheye S; BIOADAPTOR-RCT Collaborators. First randomised controlled trial comparing the sirolimus-eluting bioadaptor with the zotarolimus-eluting drug-eluting stent in patients with de novo coronary artery lesions: 12-month clinical and imaging data from the multi-centre, international, BIODAPTOR-RCT. EClinicalMedicine. 2023 Oct 24;65:102304. doi: 10.1016/j.eclinm.2023.102304. eCollection 2023 Nov. PMID 38106564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment and enrollment took place at 34 global centers including 14 in Japan and 20 in Europe between December 2020 to February 2022. A total of 445 patients with de novo coronary artery lesions were enrolled and randomly assigned to either the DynamX arm or the Resolute Onyx arm.
Period: Overall Study
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Started | 223 | 222
Completed | 221 | 215
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent | Total
Number analyzed (Participants) | 223 | 222 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.3) | 66.2 (10.1) | 66.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 174 | 173 | 347
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 110 | 113 | 223
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 0 | 0 | 0
  White | 94 | 89 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Failure (TLF)
Description: The primary endpoint of the BIOADAPTOR RCT is Target Lesion Failure (TLF), which is a composite endpoint defined as cardiac death, target-vessel MI, and Clinically-Indicated TLR
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 1.81 [.50 to 4.57] | 2.79 [1.03 to 5.97]

2. Secondary Outcome: Percentage of Participants With Target Lesion Failure (TLF)
Description: TLF is a composite endpoint defined as cardiovascular death, target-vessel MI, and Clinically-Indicated TLR
Time Frame: Through 12 months post-procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 1.8 [0.5 to 4.6] | 2.8 [1.0 to 6.0]

3. Secondary Outcome: Percentage of Participants With Patient Oriented Clinical Endpoint
Description: Overall cardiovascular outcomes from the patient's perspective. This endpoint is a composite endpoint that includes all-cause mortality (cardiac and non-cardiac), stroke, MI (target vessel and non-target vessel) and revascularization (target vessel and non-target vessel)
Time Frame: Through 12 months
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 222 | 216
percentage of participants | 6.8 [3.8 to 10.9] | 7.9 [4.7 to 12.3]

4. Secondary Outcome: Percentage of Participants With Composite of All-cause Mortality
Description: A composite of all-cause mortality, MI (target vessel or non-target vessel) and revascularization (target vessel or non-target vessel)
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 222 | 216
percentage of participants | 6.8 [3.8 to 10.9] | 7.9 [4.7 to 12.3]

5. Secondary Outcome: Percentage of Participants With Composite of Cardiovascular Death, TVMI and ID-TVR Revascularization
Description: Composite of cardiac death, target vessel myocardial infarction (TV-MI), or ischemia-driven target vessel revascularization (ID-TVR)
Time Frame: Through 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 1.8 [0.5 to 4.6] | 3.7 [1.6 to 7.2]

6. Secondary Outcome: Percentage of Participants With Cardiovascular Death, Stroke, MI and Revascularization
Description: Composite of cardiovascular death, stroke, MI (target vessel and non-target vessel) and revascularization (target vessel and non-target vessel)
Time Frame: Through 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 6.3 [3.5 to 10.4] | 7.4 [4.3 to 11.8]

7. Secondary Outcome: Percentage of Participants With Cardiovascular Death, MI and Revascularization
Description: Composite of cardiovascular death, MI (target vessel or non-target vessel) and revascularization (target vessel or non-target vessel)
Time Frame: Through 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 6.3 [3.5 to 10.4] | 7.4 [4.3 to 11.8]

8. Secondary Outcome: Percentage of Participants With Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: Number of Patients with Clinically Indicated Target Lesion Revascularization (CI-TLR)
Time Frame: Through 12 months post-procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 0.9 [0.1 to 3.2] | 0.5 [0.0 to 2.6]

9. Secondary Outcome: Percentage of Participants With Target Lesion Revascularization (TLR)
Description: Target lesion revascularization
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 1.4 [0.3 to 3.9] | 0.9 [0.1 to 3.4]

10. Secondary Outcome: Percentage of Participants With Target Vessel Revascularization (TVR)
Description: Re-PCI or CABG of the target vessel due to in-segment restenosis or other complications
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 1.4 [0.3 to 3.9] | 1.9 [0.5 to 4.7]

11. Secondary Outcome: Percentage of Participants With Clinically Indicated TVR (CI-TVR)
Description: Re-PCI or CABG in the target vessel due to restenosis or other complications
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 0.9 [0.1 to 3.2] | 1.4 [0.3 to 4.1]

12. Secondary Outcome: Percentage of Participants With Revascularization (Target Vessel or Non-target Vessel)
Description: Revascularization of the target vessel or non-target vessel due to in-segment restenosis or other complications
Time Frame: Through 12 months post procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 5.4 [2.8 to 9.3] | 5.2 [2.6 to 9.1]

13. Secondary Outcome: Percentage of Participants With Q-wave MI
Description: CK post procedure is twice the upper limit of the reference value or higher, with new pathological Q-wave on 2 or more contiguous ECG leads and if CK-MB is measured, CK-MB is positive, if no CKMB then troponin is positive.
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 0.0 [0.0 to 1.7] | 0.9 [0.1 to 3.4]

14. Secondary Outcome: Percentage of Participants With Non Q-wave MI
Description: CK post procedure is twice the upper limit of the reference value or higher, without new pathological Q-waves. If CK-MB is measured, CK-MB is positive, if no CKMB then troponin is positive.
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 0.9 [0.1 to 3.2] | 0.9 [0.1 to 3.4]

15. Secondary Outcome: Percentage of Participants With MI (Target Vessel or Non-target Vessel)
Description: MI is defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 1.4 [0.3 to 3.9] | 1.9 [0.5 to 4.7]

16. Secondary Outcome: Percentage of Participants With Target Vessel MI
Description: MI is defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 1.4 [0.3 to 3.9] | 1.9 [0.5 to 4.7]

17. Secondary Outcome: Percentage of Participants With All-cause Mortality
Description: As defined per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 222 | 216
percentage of participants | 0.5 [0.0 to 2.5] | 1.4 [0.3 to 4.0]

18. Secondary Outcome: Percentage of Participants With Cardiovascular Death
Description: As defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 0.0 [0.0 to 1.7] | 0.9 [0.1 to 3.3]

19. Secondary Outcome: Percentage of Participants With Composite of Cardiovascular Death or Target Vessel MI
Description: Target Vessel Related Death or MI
Time Frame: Through 12 months post procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 215
percentage of participants | 1.4 [0.3 to 3.9] | 2.8 [1.0 to 6.0]

20. Secondary Outcome: Percentage of Participants With Composite of All-cause Death or MI
Description: Target vessel or non-target vessel related death or MI
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 222 | 216
percentage of participants | 1.8 [0.5 to 4.5] | 3.2 [1.3 to 6.6]

21. Secondary Outcome: Percentage of Participants With Composite of All-cause Death, MI (Target Vessel or Non-target Vessel), or TVR
Description: Any Death, any MI and any Target Vessel Revascularization
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 222 | 216
percentage of participants | 2.7 [1.0 to 5.8] | 4.6 [2.2 to 8.3]

22. Secondary Outcome: Percentage of Participants With Composite of Probable or Definite Stent Thrombosis
Description: Defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 214
percentage of participants | 0.5 [0.0 to 2.5] | 0.5 [0.0 to 2.6]

23. Secondary Outcome: Percentage of Participants With Probable Stent Thrombosis
Description: Defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months post-procedure
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 214
percentage of participants | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.6]

24. Secondary Outcome: Percentage of Participants With Definite Stent Thrombosis
Description: Defined as per the Academic Research Consortium (ARC-2) criteria
Time Frame: Through 12 months
Population: The denominator reflects the number of evaluable participants for the outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
Number analyzed (Participants) | 221 | 213
percentage of participants | 0.5 [0.0 to 2.5] | 0 [0.0 to 1.7]

ADVERSE EVENTS:
Time Frame: Through 12-month post procedure
Description: Site reported AE and SAE's were reported by sites using MedDRA preferred terms. All study endpoint-related adverse events through 12 months, including death, myocardial Infarction, revascularization, stent thrombosis, and stroke, were adjudicated. All-cause mortality was calculated based off the number of evaluable participants at 12 months. Site reported SAE and AE table were calculated based on the total number of enrolled participants from the start of the trial.
Arm/Group | Elixir Bioadaptor (ELX1805J) | Medtronic Resolute Onyx Stent
All-Cause Mortality (participants affected / at risk) | 1/222 | 3/216
Serious Adverse Events (participants affected / at risk) | 60/223 | 44/222
Other Adverse Events (participants affected / at risk) | 128/223 | 124/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elixir Bioadaptor (ELX1805J) (N=223) | Medtronic Resolute Onyx Stent (N=222)
Death - Cardiovascular (Cardiac disorders) | 1 | 1
Death - Non-Cardiovascular (General disorders) | 0 | 1
MI (Cardiac disorders) | 1 | 2 — MI
Revascularization Re-PCI (Cardiac disorders) | 12 | 10
Revascularization - CABG (Cardiac disorders) | 1 | 1
Stent Thrombosis - Definite (Cardiac disorders) | 1 | 0
Stent Thrombosis - Probable (General disorders) | 0 | 0
Stent Thrombosis - Possible (General disorders) | 0 | 0
CVA - TIA (Nervous system disorders) | 0 | 0
CVA - Ischemic (Nervous system disorders) | 0 | 0
CVA - Haemorrhagic (Nervous system disorders) | 0 | 0
Bleeding (Injury, poisoning and procedural complications) | 3 | 3
Other (General disorders) | 41 | 25
Death - Unknown (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elixir Bioadaptor (ELX1805J) (N=223) | Medtronic Resolute Onyx Stent (N=222)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 5 | 5
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 3
Atrial tachycardia (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Chest discomfort (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 3 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Dyspnoea (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myopericarditis (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Thoracic pain (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Congenital spinal stenosis (Congenital, familial and genetic disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Barrett"s oesophagus (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum itestial haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Hemmorhages (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 2 | 0
Melanea (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 8 | 13
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 3
Peripheral swelling (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 2 | 0
Vascular stent thrombosis (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 8 | 13
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 5
Coronary artery dissection (Injury, poisoning and procedural complications) | 5 | 10
Coronary artery occlusion (Injury, poisoning and procedural complications) | 1 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 3
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Reperfusion injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Vessel perforation (Injury, poisoning and procedural complications) | 2 | 0
Vessel puncture site haematoma (Injury, poisoning and procedural complications) | 1 | 1
Vessel puncture site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vessel puncture site swelling (Injury, poisoning and procedural complications) | 0 | 1
Angiogram (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Magnetic resonance imaging abnormal (Investigations) | 0 | 1
Myocardial necrosis marker increased (Investigations) | 9 | 4
Prostatic specific antigen increased (Investigations) | 0 | 1
Troponin I increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Ureteroscopy (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 2
Spinal claudication (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Calculus urinary (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 2 | 2
Craniotomy (Surgical and medical procedures) | 0 | 1
Finger amputation (Surgical and medical procedures) | 1 | 0
Keratoplasty (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Skin cyst excision (Surgical and medical procedures) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute coronary syndrome (Vascular disorders) | 0 | 1
Aneurysm arteriovenous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Internal haemorrhage (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vein thrombosis (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 1
Lumbar spinal stenosis (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04192747/Prot_SAP_000.pdf